CLINICAL TRIAL: NCT03971877
Title: Detection of Colistin-resistant Isolates From Patients Admitted in Intensive Care Units and Oncohaematology Wards in the Region Nouvelle Aquitaine: Diagnostic Accuracy of the Detection Methods, Estimation of the Prevalence and Description of the Resistance Mechanisms.
Brief Title: Detection of Colistin-resistant Isolates From Patients of Intensive Care Units and Oncohaematology Wards.
Acronym: RESCO
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/45
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Colistin Resistance in Bacteria
Keywords: Colistin resistance in bacteria; Rectal swab; ICU; Oncohaematology; Gram negative bacteria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Colistin resistant isolates from rectal swabs or stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted in ICU or oncohaematology ward
  Interventions: Diagnostic Test: Rapid Polymyxin NP test

INTERVENTIONS:
Diagnostic Test: Rapid Polymyxin NP test — From rectal swabs of patients admitted in ICU and oncohaematology ward, investigators will use first a new culture medium (SuperPolymyxin) for screening the colistin resistant Gram negative and then a new rapid test (Rapid Polymyxin NP test) to confirm this resistance. These tests will be compared to the reference test of MIC (Minimal Inhibitory Concentration) determined by the broth micro-dilution (BMD) method.

SUMMARY:
The increasing use of colistin in multidrug resistant strains, as Enterobacteriaceae producing extended-spectrum β-lactamases or carbapenemases, is associated with the emergence of colistin resistant isolates. The main objective of this project is to estimate the diagnostic accuracy (sensitivity and specificity) of a new rapid detection test of colistin resistant strains (Rapid Polymyxin NP test) isolated in clinical settings.

DETAILED DESCRIPTION:
For 15 years, the prevalence of the extended-spectrum β-lactamases producing Enterobacteriaceae (ESBLE), resistant to the 3rd generation cephalosporins, has constantly increased worldwide. Since 2010 an additional threat appeared with the emergence of the bacteria resistant to carbapenems, the antibiotic of choice in case of infection due to ESBLE. To treat the infection due to these extremely resistant strains, there are still only few molecules, as the colistin. Very quickly, the colistin resistance appeared, especially a plasmid-born resistance described in December 2015 and which has already spread a lot, most probably from an animal reservoir. The control of the resistance dissemination requires reliable tools for detection of colistin resistant isolates, in particular in immunocompromised patients, as those of intensive care unit (ICU) or oncohaematology ward, that are often exposed to multidrug resistant strains. Currently, the colistin resistance is difficult to detect and that is probably why it was underestimated for a long time and has already diffuse worldwide. Some recent tests for the detection of colistin resistant isolates have been developed and tested in laboratory. They have now to be evaluated in clinical situation in order to be correctly used and interpreted. From rectal swabs of patients admitted in ICU and oncohaematology ward, investigators will use first a new culture medium (SuperPolymyxin) for screening the colistin resistant Gram negative bacteria and then a new rapid test (Rapid Polymyxin NP test) to confirm this resistance. These tests will be compared to the reference test of MIC (Minimal Inhibitory Concentration) determined by the broth micro-dilution (BMD) method. The isolates will be collected on the screening medium, during 12 months, from 4 centers (Mont de Marsan, Limoges, Dax, Bordeaux) and sent to Bordeaux University Hospital where the rapid test and the BMD method will be centralized.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years old
* patients admitted in ICU or in oncohaematology ward

Exclusion Criteria:

- Patients under protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICU or in oncohaematology ward
Sampling Method: Non-Probability Sample
Enrollment: 1934 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Rapid Polymyxin NP test | Up to 1 year after Inclusion (rectal swab or stool collection)
Specificity of Rapid Polymyxin NP test | Up to 1 year after Inclusion (rectal swab or stool collection)

SECONDARY OUTCOMES:
Prevalence rate of the colistin resistance | Up to 1 year after Inclusion (rectal swab or stool collection)
Bacterial species found resistant | Up to 1 year after Inclusion (rectal swab or stool collection)
Characterization of the various colistin resistance mechanisms | Up to 1 year after Inclusion (rectal swab or stool collection)
Identification of the genetic support of the resistance (plasmid or chromosome) | Up to 1 year after Inclusion (rectal swab or stool collection)

CONTACTS AND LOCATIONS:
Overall Officials: Paul PEREZ, MD-PhD, Study Chair — Unité de Soutien Méthodologique à la Recherche Clinique et Epidémiologique (USMR) du CHU de Bordeaux
Locations (4):
- France (4):
  - CHU de Bordeaux, Bordeaux
  - CH de Dax, Dax
  - CHU de Limoges, Limoges
  - CH de Mont de Marsan, Mont-de-Marsan